CLINICAL TRIAL: NCT05608993
Title: RELAX: Reducing Length of Antibiotics for Children With Ear Infections
Acronym: RELAX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Vanderbilt University Medical Center (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-1528; 1R01HS029153-01 (AHRQ)
Record Dates: First submitted 2022-10-24; First posted 2022-11-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Acute Otitis Media; Pediatric Infectious Disease; Ear Infection
Keywords: Acute Otitis Media; Ear Infections; Pediatric Infectious Disease; Electronic Health Record; Antibiotic Stewardship
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity (Experimental): Community-based clinics and/or urgent care centers that are assigned to the high intensity arm will receive the high intensity intervention.
  Interventions: Other: High Intensity Intervention
- Low Intensity (Experimental): Community-based clinics and/or urgent care centers that are assigned to the low intensity arm will receive the low intensity intervention.
  Interventions: Other: Low Intensity Intervention

INTERVENTIONS:
Other: High Intensity Intervention — The High Intensity intervention will include clinician education, individualized clinician audit and feedback with peer comparison, and electronic health record (EHR) changes of prescription fields.
  Arms: High Intensity
Other: Low Intensity Intervention — The Low Intensity intervention will include clinician education and EHR changes only.
  Arms: Low Intensity

SUMMARY:
The overarching goal of this study is to evaluate the effectiveness and implementation outcomes of two low-cost interventions of different intensities to increase prescribing of recommended short antibiotic durations for acute otitis media (AOM) for children 2 years of age and older. A multi-center cluster randomized controlled trial using a hybrid type 2 implementation effectiveness design will be used to evaluate interventions. The High-Intensity intervention will include clinician education, individualized clinician audit and feedback with peer comparison, and electronic health record (EHR) changes of prescription fields, whereas the Low-Intensity intervention will include clinician education and EHR changes. In total, 46 community-based clinics and/or urgent care centers across two distinct geographic regions in the United States will be randomized to one of the two interventions. The Practical Robust Implementation and Sustainability Model (PRISM) will be used to guide implementation and the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework will be used to evaluate outcomes. A mixed-methods approach will be used in the pre-implementation and evaluation phases and will utilize quantitative analyses, semi-structured interviews, focus groups, surveys, and cost analyses. National stakeholders at the American Academy of Pediatrics and the Centers for Disease Control and Prevention will assist with dissemination of findings and scaling of interventions.

DETAILED DESCRIPTION:
Acute otitis media (AOM) is the most commonly cited indication for antibiotics in children, accounting for 24% of all pediatric antibiotic prescriptions and affecting 60% of children by 3 years of age. For most children ≥ 2 years of age with AOM, 5-7 days, rather than 10 days, of antibiotics have been shown to be sufficient and result in fewer adverse drug events with similar failure and recurrence rates. Thus, national guidelines recommend short durations of antibiotics for non-severe AOM in this age group. Despite these recommendations, >94% of children ≥2 years of age are prescribed longer than recommended antibiotic durations and over 41% of antibiotic exposure days for AOM in this age group are likely unnecessary. In a recent pilot study that compared a low-cost High-intensity intervention with clinician education, individualized clinician audit and feedback with peer comparison and electronic health record (EHR) changes of prescription fields to a Low-intensity intervention with only EHR changes prescribing of recommended short antibiotic durations increased significantly (76% and 50%, absolute percentage). A definite study is needed to make appropriate recommendations on which intervention to implement, while minimizing resource utilization.

The overarching goal of this study is to evaluate the effectiveness and implementation outcomes of two low-cost pragmatic interventions of different intensities to increase prescribing of recommended short antibiotic durations for AOM for children 2 years of age and older. A multi-center cluster randomized controlled trial using a hybrid type 2 implementation effectiveness design will be used to evaluate interventions. The High-intensity intervention will include clinician education, individualized clinician audit and feedback with peer comparison, and EHR changes of prescription fields, whereas the Low-intensity intervention will include clinician education and EHR changes. In total, 46 community-based clinics and/or urgent care centers across two distinct geographic regions in the United States will be randomized to one of the two interventions. The Practical Robust Implementation and Sustainability Model will be used to guide implementation and the Reach Effectiveness Adoption Implementation Maintenance framework will be used to evaluate outcomes. A mixed-methods approach will be used in the pre-implementation and evaluation phases and will utilize quantitative analyses, semi-structured interviews, focus groups, surveys, and cost analyses.

ELIGIBILITY:
Inclusion Criteria:

A. Secondary use data of encounters for children with AOM

1. Aged 2-17-years-old (inclusive)
2. Diagnosis of AOM by ICD10 code
3. AOM is uncomplicated
4. Prescribed an oral antibiotic

B. Clinician and administrator interviews

1. Licensed clinician (physician or advanced practice clinician) that cares for children with AOM
2. Practices in an intervention study site
3. Is not a medical trainee (student, resident, fellow, etc.)
4. Aged >=18 years-no maximum

C. Parent focus groups

1. Parent or legal guardian of a child aged 2-17 years that has had AOM diagnosed at Vanderbilt University Medical Center or Washington University
2. 18 years of age or older and able/willing to consent

D. Clinician and administrator surveys

1. Licensed clinician (physician or advanced practice clinician) that cares for children with AOM
2. Practices in an intervention study site
3. Is not a medical trainee (student, resident, fellow, etc.)
4. Aged >=18 years-no maximum

Exclusion Criteria:

A. Secondary use data of encounters for children with AOM

1. Complicated infection (determined a priori)

B. Clinician and administrator interviews 1. Medical trainee

C. Parent focus groups

1. Not parent or legal guardian
2. Does not speak English or Spanish (focus groups can only be conducted in these languages).

D. Clinician and administrator surveys

1. Medical trainee

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of children ≥ 2 years of age with AOM that are prescribed a short duration (5 days) of antibiotics. | 5 years
  Determine the effectiveness of a High and Low intensity intervention to increase prescribing of recommended antibiotic durations (short, 5 days) for AOM in children ≥ 2 years of age.

SECONDARY OUTCOMES:
Mean days of antibiotics prescribed | 5 years
  Mean number of days of antibiotics prescribed for children ≥ 2 years of age with AOM
Adverse drug event | 5 years
  Number of adverse drug events among children ≥ 2 years of age prescribed antibiotics for AOM
Treatment failure | 5 years
  Treatment failure defined as a new antibiotic associated with an AOM encounter within 3-14 days of the initial encounter.
Recurrence | 5 years
  Recurrence defined as a new antibiotic associated with an AOM encounter within 15-30 days of initial encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Holly M Frost, MD, Principal Investigator — Intermountain Health Care, Inc.; Sophie E Katz, MD, Principal Investigator — Vanderbilt University Medical Center; Jason Newland, MD, Principal Investigator — Washington University School of Medicine; Timothy C Jenkins, MD, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Rinehart DJ, Gilbert A, O'Leary S, Katz SE, Frost HM. Reducing antibiotic duration for acute otitis media: clinician, administrator, and parental insights to inform implementation of system-level interventions. Antimicrob Steward Healthc Epidemiol. 2025 Jan 6;5(1):e3. doi: 10.1017/ash.2024.469. eCollection 2025. PMID 39781291
- [Derived] Keith A, Jenkins TC, O'Leary S, Stein AB, Katz SE, Newland J, Rinehart DJ, Gilbert A, Dodd S, Terrill CM, Frost HM. Reducing length of antibiotics for children with ear infections: protocol for a cluster-randomized trial in the USA. J Comp Eff Res. 2023 Nov;12(11):e230088. doi: 10.57264/cer-2023-0088. Epub 2023 Oct 19. PMID 37855227